CLINICAL TRIAL: NCT02581007
Title: Reduced Intensity Conditioning and Transplantation of Partially HLA-Mismatched Peripheral Blood Stem Cells for Patients With Hematologic Malignancies
Brief Title: Reduced Intensity Conditioning Transplant Using Haploidentical Donors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northside Hospital, Inc. (Other)
Collaborators: Blood and Marrow Transplant Group of Georgia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSH 1132
Record Dates: First submitted 2015-10-16; First posted 2015-10-20 (Estimated); Results first posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Chronic Myelogenous Leukemia; Acute Myelogenous Leukemia; Myelodysplastic Syndrome; Acute Lymphocytic Leukemia; Chronic Lymphocytic Leukemia; Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma; Myelofibrosis; CMML; Multiple Myeloma
Keywords: CML; AML; MDS; ALL; CLL/CPL; HD; NHL; MPS; CMML; MM
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Hodgkin Disease; Lymphoma, Non-Hodgkin; Primary Myelofibrosis; Multiple Myeloma | interventions — fludarabine; fludarabine phosphate; Melphalan; Cyclophosphamide; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reduced-Intensity Mismatched Transplant (Experimental): Fludarabine, Melphalan & Post-transplant cyclophosphamide
  Interventions: Drug: Fludarabine; Drug: Melphalan; Drug: Cyclophosphamide; Procedure: peripheral blood stem cell transplant

INTERVENTIONS:
Drug: Fludarabine — fludarabine (30mg/m2) given every day starting on Day -6 through Day -2;
  Other Names: Fludara
Drug: Melphalan
  Other Names: melphalan (140mg/m2) given one time on Day -1.
Drug: Cyclophosphamide — cyclophosphamide (50mg/kg) given every day starting on Day 3 through Day 4.
  Other Names: Cytoxan
Procedure: peripheral blood stem cell transplant
  Other Names: HSCT

SUMMARY:
This trial will evaluate the safety and efficacy of a reduced intensity allogeneic HSCT from partially HLA-mismatched first-degree relatives utilizing PBSC as the stem cell source. The primary objective of the study is to estimate the incidence of graft rejection and acute GVHD. A secondary objective will be to estimate the incidence of the relapse, NRM, OS, chronic GVHD and EFS.

DETAILED DESCRIPTION:
Patients will receive a haploidentical transpalnt using a fludarabine melphalan prepartive regimen. Patients will get cyclophosphamide on days 3 & 4 post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* No available matched related or unrelated donor, OR a matched related or unrelated donor will not be available in time frame necessary to perform potentially curative transplant
* Availability of 3/6 - 5/6 matched (HLA-A, B, DR) related donor (donor must have negative HLA cross-match in host vs. graft direction)
* Karnofsky status ≥70%
* One of the following high-risk malignancies:

  1. Chronic Myelogenous Leukemia: Chronic myelogenous leukemia in chronic phase, resistant or intolerant to available tyrosine kinase inhibitors; Chronic myelogenous leukemia in accelerated phase; Chronic myelogenous leukemia with blast crisis that has entered into a second chronic phase following induction chemotherapy
  2. Acute Myelogenous Leukemia in first or greater remission
  3. Myelodysplastic Syndrome at least one of the following: treatment-related; monosmy 7, complex cytogenetics or other high risk karyotype; IPSS score of 1.0 or greater; neutropenia or cytopenia requiring transfusion not responding to therapy; peripheral or BM blast count of <10%; CMML
  4. Acute lymphocytic leukemia/lymphoblastic lymphoma: 2nd or subsequent complete remission; first complete remission; marrow blasts <5%, but persistence of minimal residual disease by flow cytometry, cytogenetics, or FISH
  5. Chronic Lymphocytic Leukemia/Prolymphocytic Leukemia: previously treated disease that has either relapsed or failed to respond adequately to conventional-dose therapy including purine analogs
  6. Hodgkin's or Non-Hodgkin's Lymphoma (including low-grade, mantle cell, and intermediate-grade/diffuse): previously treated disease that has either relapsed or failed to respond adequately to conventional-dose therapy or autologous transplantation
  7. Myeloproliferative diseases (myelofibrosis, CMML)
  8. Multiple Myeloma with relapse after a prior autologous transplant or eligible for allogeneic HSCT based on other risk factors

Exclusion Criteria:

* not be excluded on basis of sex, racial, or ethnic backgrounds
* poor cardiac function: left ventricular ejection fraction <40%
* poor pulmonary function: FEV1 and FVC <50% predicted
* poor liver function: bilirubin >2 mg/dl (not due to hemolysis, Gilbert's or primary malignancy)
* poor renal function: Creatinine >2.0mg/dl or creatinine clearance (calculated creatinine clearance is permitted) < 40 mL/min based on Traditional Cockcroft-Gault formula: 140 - age (yrs) x Smaller of Actual Weight vs. Ideal Body Weight (kg) / 72 x Serum creatinine (mg/dl)
* HIV-positive
* prior allogeneic transplant
* women of childbearing potential who currently are pregnant or who are not practicing adequate contraception
* any debilitating medical or psychiatric illness which would preclude their giving informed consent or their receiving optimal treatment and follow-up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-10-26 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2020-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melhem Solh, MD, Principal Investigator — Northside Hospital
Locations (1):
- Northside Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szydlo R, Goldman JM, Klein JP, Gale RP, Ash RC, Bach FH, Bradley BA, Casper JT, Flomenberg N, Gajewski JL, Gluckman E, Henslee-Downey PJ, Hows JM, Jacobsen N, Kolb HJ, Lowenberg B, Masaoka T, Rowlings PA, Sondel PM, van Bekkum DW, van Rood JJ, Vowels MR, Zhang MJ, Horowitz MM. Results of allogeneic bone marrow transplants for leukemia using donors other than HLA-identical siblings. J Clin Oncol. 1997 May;15(5):1767-77. doi: 10.1200/JCO.1997.15.5.1767. PMID 9164184
- [Background] Anasetti C, Amos D, Beatty PG, Appelbaum FR, Bensinger W, Buckner CD, Clift R, Doney K, Martin PJ, Mickelson E, et al. Effect of HLA compatibility on engraftment of bone marrow transplants in patients with leukemia or lymphoma. N Engl J Med. 1989 Jan 26;320(4):197-204. doi: 10.1056/NEJM198901263200401. PMID 2643045
- [Background] Kernan NA, Flomenberg N, Dupont B, O'Reilly RJ. Graft rejection in recipients of T-cell-depleted HLA-nonidentical marrow transplants for leukemia. Identification of host-derived antidonor allocytotoxic T lymphocytes. Transplantation. 1987 Jun;43(6):842-7. PMID 3296349
- [Background] Aversa F, Terenzi A, Tabilio A, Falzetti F, Carotti A, Ballanti S, Felicini R, Falcinelli F, Velardi A, Ruggeri L, Aloisi T, Saab JP, Santucci A, Perruccio K, Martelli MP, Mecucci C, Reisner Y, Martelli MF. Full haplotype-mismatched hematopoietic stem-cell transplantation: a phase II study in patients with acute leukemia at high risk of relapse. J Clin Oncol. 2005 May 20;23(15):3447-54. doi: 10.1200/JCO.2005.09.117. Epub 2005 Mar 7. PMID 15753458
- [Background] Bashey A, Solomon SR. T-cell replete haploidentical donor transplantation using post-transplant CY: an emerging standard-of-care option for patients who lack an HLA-identical sibling donor. Bone Marrow Transplant. 2014 Aug;49(8):999-1008. doi: 10.1038/bmt.2014.62. Epub 2014 May 19. PMID 24842530
- [Background] O'Donnell PV, Luznik L, Jones RJ, Vogelsang GB, Leffell MS, Phelps M, Rhubart P, Cowan K, Piantados S, Fuchs EJ. Nonmyeloablative bone marrow transplantation from partially HLA-mismatched related donors using posttransplantation cyclophosphamide. Biol Blood Marrow Transplant. 2002;8(7):377-86. doi: 10.1053/bbmt.2002.v8.pm12171484.
- [Background] Solomon SR, Sizemore CA, Sanacore M, Zhang X, Brown S, Holland HK, Morris LE, Bashey A. Haploidentical transplantation using T cell replete peripheral blood stem cells and myeloablative conditioning in patients with high-risk hematologic malignancies who lack conventional donors is well tolerated and produces excellent relapse-free survival: results of a prospective phase II trial. Biol Blood Marrow Transplant. 2012 Dec;18(12):1859-66. doi: 10.1016/j.bbmt.2012.06.019. Epub 2012 Aug 1. PMID 22863841
- [Background] Solomon SR, Sizemore CA, Sanacore M, Zhang X, Brown S, Holland HK, Morris LE, Bashey A. Total Body Irradiation-Based Myeloablative Haploidentical Stem Cell Transplantation Is a Safe and Effective Alternative to Unrelated Donor Transplantation in Patients Without Matched Sibling Donors. Biol Blood Marrow Transplant. 2015 Jul;21(7):1299-307. doi: 10.1016/j.bbmt.2015.03.003. Epub 2015 Mar 19. PMID 25797174

RESULTS

PARTICIPANT FLOW:
Groups:
- Reduced-Intensity Mismatched Transplant: Fludarabine, Melphalan & Post-transplant cyclophosphamide
  Fludarabine: fludarabine (30mg/m2) given every day starting on Day -6 through Day -2;
  Melphalan
  Cyclophosphamide: cyclophosphamide (50mg/kg) given every day starting on Day 3 through Day 4.
  peripheral blood stem cell transplant
Period: Overall Study
Arm/Group | Reduced-Intensity Mismatched Transplant
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Reduced-Intensity Mismatched Transplant
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: years] | 57 [35 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Graft Rejection
Description: Measurement of donor cells vs. recipient cells
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced-Intensity Mismatched Transplant
Number analyzed (Participants) | 25
Participants | 3

2. Secondary Outcome: Overall Survival
Description: Number of participants still alive 2 years after transplant
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Reduced-Intensity Mismatched Transplant
Number analyzed (Participants) | 25
percentage of patients
  1 yr post-transplant | 68 [46 to 82]
  2 yr post-transplant | 56 [33 to 74]

3. Secondary Outcome: Relapse Incidence
Description: Number of patients with disease reoccurrence at 1 and 2 years post-transplant
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Reduced-Intensity Mismatched Transplant
Number analyzed (Participants) | 25
percentage of patients
  1 yr post-transplant | 24 [10 to 42]
  2 yr post-transplant | 36 [17 to 55]

4. Secondary Outcome: GVHD Incidence
Description: The number of participants that developed graft-versus-host-disease before or at 100 days after transplant
Time Frame: 100 days
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Reduced-Intensity Mismatched Transplant
Number analyzed (Participants) | 25
percentage of patients
  Grades II to IV acute GVHD | 20 [8 to 37]
  Grades III to IV acute GVHD | 8 [2 to 22]
  Moderate chronic GVHD | 16 [5 to 33]
  Severe chronic GVHD | 12 [3 to 27]

ADVERSE EVENTS:
Time Frame: 100 days for adverse events, overall survival over 2 years
Arm/Group | Reduced-Intensity Mismatched Transplant
All-Cause Mortality (participants affected / at risk) | 3/25
Serious Adverse Events (participants affected / at risk) | 23/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Reduced-Intensity Mismatched Transplant (N=25)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
confusion (Nervous system disorders) | 2
sepsis (Infections and infestations) | 4
renal failure (Renal and urinary disorders) | 1
hypoxia (Respiratory, thoracic and mediastinal disorders) | 7
pericardial effusion (Cardiac disorders) | 3
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3
sinusitis (Infections and infestations) | 1
esophagitis (Gastrointestinal disorders) | 2
chest pain (General disorders) | 1
mucositis (Gastrointestinal disorders) | 1
tachycardia (Cardiac disorders) | 1
elevated liver enzymes (Metabolism and nutrition disorders) | 1
fever (General disorders) | 15
hallucinations (Psychiatric disorders) | 1
cardiac arrest (Cardiac disorders) | 1
anorexia (Gastrointestinal disorders) | 1
graft-versus-host-disease (Immune system disorders) | 1
pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
bacteremia infection (Infections and infestations) | 6
nausea (Gastrointestinal disorders) | 4
vomiting (Gastrointestinal disorders) | 4
diarrhea (Gastrointestinal disorders) | 4
superficial venous thrombosis (Cardiac disorders) | 1
hypotension (Cardiac disorders) | 1
hypertension (Cardiac disorders) | 1
thrombocytopenia (Investigations) | 3
deep venous thrombosis (Cardiac disorders) | 1
tumor lysis syndrome (Metabolism and nutrition disorders) | 1
cytokine release syndrome (Immune system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Reduced-Intensity Mismatched Transplant (N=25)
leukopenia (Investigations) | 25
neutropenia (Investigations) | 25
BK virus (Renal and urinary disorders) | 2
anemia (Investigations) | 10
rash (Skin and subcutaneous tissue disorders) | 4
hypokalemia (Metabolism and nutrition disorders) | 3
hyponatremia (Metabolism and nutrition disorders) | 1
weight loss (Gastrointestinal disorders) | 1
syncope (Nervous system disorders) | 1
hypocalcemia (Metabolism and nutrition disorders) | 2
elevated liver enzymes (Metabolism and nutrition disorders) | 8
hypertension (Cardiac disorders) | 3
thrombocytopenia (Investigations) | 25
urinary tract infection (Renal and urinary disorders) | 1
hyperglycemia (Metabolism and nutrition disorders) | 3
hypomagnesemia (Metabolism and nutrition disorders) | 1
hypermagnesemia (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT02581007/Prot_SAP_000.pdf